CLINICAL TRIAL: NCT04487418
Title: Evaluation of the Effects of High-level Laser and Electro-cautery in Lingual Frenotomy Surgeries in Infants - Blinded Randomized Controlled Clinical Study
Brief Title: Evaluation of the Effects of High-level Laser and Electro-cautery in Lingual Frenotomy Surgeries in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lingualfrenotomy
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Lingual Frenum; High Power Laser; Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery group with electro cautery (Experimental): Surgery will be performed with electro cautery.
  Interventions: Procedure: Electro cautery surgery
- High level diode laser surgery (Experimental): High power diode laser surgery will be performed.
  Interventions: Procedure: High power diode laser surgery

INTERVENTIONS:
Procedure: Electro cautery surgery — Pre-anesthetics with therapeutic topic (benzocaine) will be administered and, as an anesthetic, or use of anesthetic drops (benzocaine or tetracaine) or local infiltrative anesthesia (2% lidocaine 1: 100,000 with adrenaline).
  The surgery will be carried out with cauterization for incision of the lingual brake, division of the brake fibers and release, removing the brake fibers that are stored in the anterior ventral free parts of the tongue until reaching the base of the tongue, which are removed or cleaned, lingual movement, and the anterior axis of the tongue is repositioned or lingual brake in that region. No sutures will be performed and should be oriented on the formation of a pseudo-membranous repair plate in the second intention that will be formed between the first and the third day after surgery.
  Postoperative care:
  Guidance will be given to the person responsible for not bringing objects to the mouth that may hurt.
  Arms: Surgery group with electro cautery
Procedure: High power diode laser surgery — Pre-anesthetics with therapeutic topic (benzocaine) and as anesthetic or use of anesthetic eye drops (benzocaine or tetracaine) or local infiltrative anesthesia (2% lidocaine 1: 100,000 with adrenaline) will be administered. The surgery will be performed with a high power diode laser (TW Surgical, MMOptics - São Carlos - Brazil). 808 nm wavelength, which can be operated in continuous or interrupted mode. Wattages from 1 to 1.5 W, up to a maximum of 2 W, can be used and must carefully respect the histological characteristics of the target tissue and the signs of overheating and carbonization, so that the choice of parameters is dynamic and very dependent on experience, mastery and care for the operator.
  Preoperative care: Guidance will be given to the person responsible for not bringing objects to the mouth that may hurt.
  Arms: High level diode laser surgery

SUMMARY:
Ankyloglossia is an anomaly that is characterized by an abnormally short, thick or thin lingual frenulum that can restrict the movements of the tongue and has been identified as one of the factors that can negatively interfere with breastfeeding, decreasing the ability of the newborn to make a clamp proper. According to the Ministry of Health in Brazil, the percentage of newborns who present this anomaly is 3% to 16%. The objective of the study will be to evaluate the release of the lingual frenulum through the lingual frenotomy performed with a high level diode laser or with an electro cautery. Methods: The present study will be a blind randomized controlled clinical trial, in which 56 volunteers, infants aged 0 to 3 months, with normal health status, who are breastfeeding, diagnosed with ankyloglossia and indication for surgery, will do lingual frenotomy. Those responsible for the children will be informed about the study procedures and after signing the Free and Informed Consent Form, authorizing them to participate in the study. The non-blinded researcher will conduct the evaluation, screening and procedures, and another blinded researcher will be the evaluator 15 days after the procedure. The distribution of volunteers in the groups will be random and randomized: Surgery Group with electro cautery (G1- EC) and Surgery Group with high power diode laser (G2-L). The procedures for patient preparation, asepsis and infection control will be strictly followed in accordance with biosafety rules. In both groups the infants will be submitted to anamnesis, clinical evaluation and standardized photograph of the lingual frenulum region before the surgical procedure and application of the Bristol frenulum evaluation protocol, the nursing mother will be submitted to the evaluation of the VAS of pain during breastfeeding, before, shortly after and 15 days after the surgical procedure for the evaluation of the result of the lingual frenotomy. Discussion: Ankyloglossia can negatively impact breastfeeding. The lingual frenotomy procedure can be performed using various surgical techniques. The use of high-power laser for this purpose has been identified as an effective resource in the incision of the lingual frenulum, with advantages in the trans-operative period, less bleeding and better visualization of the surgical field, and in the post-operative period, with reduction of edema, pain and inflammation, quality of tissue repair and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 3 months old
* Infants born within normal health standards
* Infants who are breastfeeding
* Have a diagnosis of ankyloglossia with a score of 0 to 4 according to the Bristol protocol, performed by a Speech Therapist and / or Dental Surgeon and / or Pediatrician.

Exclusion Criteria:

* Infants with changes:
* Congenital and systemic
* Blood dyscrasias
* Hemophilia, diabetes
* Nutritional weaknesses
* Imunodeficiencies
* Changes in the oral cavity
* Infants who are under medical treatment
* Use of medication
* Do not be well on the day of the surgical procedure.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2020-09-03 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-03 (Estimated)

PRIMARY OUTCOMES:
Photograph of the lingual brake region | 10 minutes
  An intraoral photograph will be performed on the planes: frontal, median sagittal of the patient, parallel to the vertical edges and occlusal to the horizontal edges with the focus on the lingual brake region. The evaluation will be performed after the surgical procedure, and after 15 days.
BRISOL | 15 minutes
  The baby will be placed on the lap of one of the guardians, adult, in the supine position, who in turn is lying in the dental chair, in some situations the knee-to-knee position may be used, and the professional should assess which will be more convenient for stabilization. protective of the patient.
  asepsis and infection control for the patient, will be strictly followed in accordance with Biosafety rules.
  In the Bristol protocol we will have a final score based on 4 points to observe: appearance of the tip of the tongue, fixation of the brake in the lower alveolus, elevation of the tongue during crying and protrusion of the tongue on the gums The evaluation will be carried out immediately after the surgery and after 15 days.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 10 minutes
  The application of the VAS pain scale will be applied to the nursing mother during breastfeeding before, shortly after and 15 days after the surgical procedure. During breastfeeding, the nursing mother will be asked about the pain in the breasts, and she must report the pain by looking at the scale mentioned, from 0 to 10 and choose the number that most relates to breast pain.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Mazzoni A, Navarro RS, Fernandes KPS, Horliana ACRT, Mesquita-Ferrari RA, Motta PB, Silva T, Gomes AO, Martimbianco ALC, Sobral APT, Santos EM, Motta LJ, Bussadori SK. Evaluation of the effects of high-level laser and electrocautery in lingual frenectomy surgeries in infants: protocol for a blinded randomised controlled clinical trial. BMJ Open. 2021 Nov 30;11(11):e050733. doi: 10.1136/bmjopen-2021-050733. PMID 34848514